CLINICAL TRIAL: NCT06217705
Title: Testing the Effects of Project Calm in Ukrainian Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: John Weisz (Unknown)
Responsible Party: Principal Investigator, John Weisz, Professor, Harvard University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB23-1653
Record Dates: First submitted 2024-01-12; First posted 2024-01-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Trauma; Anxiety; Depression; Child Behavior
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders; Depression; Child Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the intervention condition (Project Calm) immediately or after two months. Participants in the delayed Calm condition will complete a typical school activity instead (i.e., treatment as usual). All participants will complete survey measures online at baseline, immediately after receiving the intervention, and 1-, 2, 3-, and 4-months after baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be completed independently by participants online. Investigators will be blinded to condition throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Calm (Experimental): Project Calm is a ~30-minute self-guided digital intervention designed to teach children and adolescents empirically supported emotion regulation skills to facilitate self-calming when faced with intense negative emotions. Project Calm uses vignettes, interactive activities, and engaging graphics to teach youth calming skills.
  Interventions: Behavioral: Project Calm
- Delayed Receipt of Project Calm Control Condition (Other): No intervention for first two months; will receive Project Calm after 2-months and become a second-wave intervention condition.
  Interventions: Behavioral: Project Calm

INTERVENTIONS:
Behavioral: Project Calm — Project Calm is a ~30-minute self-guided digital intervention designed to teach children and adolescents empirically supported emotion regulation skills to facilitate self-calming when faced with intense negative emotions. Project Calm uses vignettes, interactive activities, and engaging graphics to teach youth calming skills.

SUMMARY:
The purpose of this study is to test the effectiveness of a universal, digital, single-session intervention for youth mental health, functioning, and well-being, when implemented with Ukrainian children and adolescents. The intervention teaches well-established procedures that research has shown to be effective in helping American children calm themselves and regulate emotions, including slowed breathing and peaceful mental imagery. The intervention has not been tested previously with Ukrainian students. Participants will be provided access to this brief online program as part of the school curriculum. Students will be randomly assigned to receive the digital program either immediately or after 2 months. This 2-month lag will allow for evaluating the effectiveness of Project Calm in improving students' mental health, well-being, and self-calming skills. This will also allow for evaluating the effectiveness of such an intervention for war-exposed youths for whom these interventions may be especially helpful given the gap between these children's needs for mental health services and the very limited availability of clinicians

DETAILED DESCRIPTION:
Russia's invasion of Ukraine has deeply impacted the nation's children, perhaps most strikingly those who remain in Ukraine and are confronted by the trauma of war. 2.5 million have fled their homes, but even those still at home endure explosions, violence, loss of loved ones, and an estimated average of 900 hours hiding in bunkers. Research in Ukraine shows high levels of child mental health (MH) problems, including anxiety, depression, interpersonal stress, and difficulty regulating emotions. PI Weisz works with child MH researchers and clinicians from Ukraine and 5 other countries (the GROW consortium) to plan psychological support for these children. The group has concluded that Ukrainian-language digital MH interventions teaching evidence-based coping skills are the optimum form of early psychological support at this time, given the massive number of war-exposed Ukrainian children, the dearth of professional clinicians, and the ready accessibility of digital devices. Brief digital interventions (BDIs) for MH have been found effective with children in >90 randomized controlled trials (RCTs). They require no professional training or funding, and are easily implemented via digital devices used in nearly all schools. Ukrainian children may be helped via a BDI that teaches them evidence-based procedures for calming themselves when they experience distressing emotions.

The Harvard Lab for Youth Mental Health is collaborating with Ukrainian schools in the Zhytomyr region, which has been repeatedly targeted by Russian missiles since the first month of the invasion, spreading fear throughout the population and destroying airports, residential neighborhoods, hospitals, and at least one school. Children in Zhytomyr experience war-related MH problems identified in Ukrainian research reviews, including anxiety, sadness, and difficulty calming and regulating distressing negative emotions. Students will be offered a BDI that addresses these problems by teaching well-established skills that have robust empirical support: Project Calm teaches children to calm and regulate distressing emotions by using skills such as slowed breathing, relaxing of tense muscles, and peaceful mental imagery. This 30-minute BDI, which has been refined via student and school staff feedback over a 2-year period, is highly rated by children and teens, and has already been accessed >1000 times in North America.

Project Calm will be tested via an RCT with a time-matched, school-related control activity; students will be randomized 50/50 to complete Project Calm after the baseline assessment or after a 2-month lag. Students in grades 4-12 will complete MH, wellbeing, and BDI-skills measures at baseline and 1-, 2-, 3-, and 4-months post-baseline. Data collection will span January - June of 2024. Findings may point the way to a highly scalable, accessible, and disseminable approach to MH support-easily implemented in schools or community settings-that could benefit Ukrainian children and, with translation and adaptation, war-affected children of other nations.

ELIGIBILITY:
Inclusion Criteria:

* Youth in grades 4+ at partnering schools for Ukrainian children
* Youth and at least one guardian consent to adolescent participation in study
* Youth reads Ukrainian well enough to effectively complete the digital programs
* Youth has access to a digital device

Exclusion Criteria:

* Youth does not have access to a digital device
* Youth has an intellectual disability that precludes comprehension of the program content

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 728 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Behavior and Feelings Survey (Internalizing Subscale) | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Perceived Program Acceptability and Helpfulness | Assessed immediately post-intervention
  Post-intervention feedback on the program's perceived acceptability and helpfulness as measured via a 7-item measure, with each item rated on a 1-5 scale, with higher scores indicating greater acceptability and helpfulness.

SECONDARY OUTCOMES:
Change in Behavior and Feelings Survey (Externalizing Subscale) | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Emotion Regulation Mechanisms of Change Questions | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups
  Emotion Regulation Mechanisms of Change Questions - Assessed at all time points via a novel 3-item measure (0-10 scale) evaluating participants' calming skills. Specific items include:
  * When I feel tense or nervous, I can calm myself.
  * When I feel scared, I can calm myself.
  * When I feel angry, I can calm myself.
Youth Top Problems | Assessed at baseline
  Assessed via the Youth Top Problems Assessment (Herren et al., 2018). Items are rated on a scale from 0 (not a problem at all) to 4 (a very big problem).
Peabody Treatment Progress Battery's Life Satisfaction Scale | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups
  Assessed via the Peabody Treatment Progress Battery's Life Satisfaction Scale. Items are rated on a scale from 1 (very dissatisfied) to 5 (very satisfied).
Treatment Expectancy Questions | Assessed immediately pre-intervention
  Treatment expectations will be assessed at pre-intervention via a novel 4-item measure (0-10 scale) evaluating participants' expectations of intervention effects.
Sensitivity | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups
  Assessed at all time points via the Highly Sensitive Person Scale (Baryla-Matejczuk et al., 2022). Items are rated on a scale from 1 (not at all) to 7 (definitely).
Trauma Symptoms | Assessed at baseline, 1-month, 2-month, 3-month, and 4-month follow-ups]
  Assessed at all time points via the Short Post-Traumatic Stress Disorder Rating Interview (SPRINT-10; Connor & Davidson, 2001). Items are rated on a scale from 0 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Analytic code will be made available upon publication of trial results. Study protocol and statistical plan are available on Open Science Framework.

REFERENCES:
- [Derived] Steinberg JS, Sun J, Venturo-Conerly KE, Sood G, Mair P, Davydenko O, Porzak R, Ougrin D, Weisz JR. Randomized trial testing a self-guided digital mental health intervention teaching calming skills for Ukrainian children. Npj Ment Health Res. 2025 May 16;4(1):20. doi: 10.1038/s44184-025-00134-w. PMID 40379908